CLINICAL TRIAL: NCT01074047
Title: A Phase 3, Multicenter, Randomized, Open-Label, Study of Azacitidine (Vidaza®) Versus Conventional Care Regimens for the Treatment of Older Subjects With Newly Diagnosed Acute Myeloid Leukemia
Brief Title: Study of Vidaza Versus Conventional Care Regimens for the Treatment of Acute Myeloid Leukemia (AML)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZA-AML-001
Record Dates: First submitted 2010-02-16; First posted 2010-02-24 (Estimated); Results first posted 2015-02-26 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Cytarabine; Vidaza; azacitidine; Intensive Chemotherapy; Low Dose Cytarabine; Celgene
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azacitidine (Experimental): Azacitidine daily for 7 days for 28 day cycles until disease progression or unacceptable toxicity
  Interventions: Drug: Azacitidine
- Conventional Care Regimen (Active Comparator): Conventional Care Regimen
  Interventions: Drug: Conventional Care Regimen

INTERVENTIONS:
Drug: Azacitidine — 75 mg/m^2 subcutaneous (SC) daily for 7 days for 28 day cycles until disease progression or unacceptable toxicity
  Other Names: Vidaza
  Arms: Azacitidine
Drug: Conventional Care Regimen — Physician pre-selects prior to randomization from one of the following:
  * Intensive chemotherapy (cytarabine 100-200 mg/m^2 continuous intravenous infusion for 7 days + anthracycline IV x 3 days) + Best Supportive Care; induction with up to 2 consolidation cycles
  * Low-dose cytarabine 20 mg subcutaneous (SC) twice a day (BID) for 10 days, for 28 day cycles + BSC; until disease progression or unacceptable toxicity
  * Best Supportive Care only; until study end
  Arms: Conventional Care Regimen

SUMMARY:
The purpose of this study is to compare the effect of azacitidine (Vidaza) to conventional care regimens on overall survival in elderly AML patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following

  * Newly diagnosed de novo acute myeloid leukemia (AML)
  * AML secondary to myelodysplastic syndromes (MDS)
  * AML secondary to exposure to leukemogenic therapy or agents with primary malignancy in remission for at least 2 years
* Bone marrow blasts >30%
* Age ≥ 65 years
* Easter Cooperative Oncology Group (ECOG) 0-2

Exclusion Criteria:

* Previous cytotoxic or biologic treatment for AML (except hydroxyurea)
* Previous treatment with azacitidine, decitabine or cytarabine
* Prior use of targeted therapy agents (e.g., FLT3 inhibitors, other kinase inhibitors)
* AML French American British subtype (FAB M3)
* AML associated with inv(16), t(8;21), t(16;16), t(15:17), or t(9;22) karyotypes
* Prior bone marrow or stem cell transplantation
* Candidate for allogeneic bone marrow or stem cell transplant
* Diagnosis of malignant disease within the previous 12 months (excluding base cell carcinoma, "in-situ" carcinoma of the cervix or breast or other local malignancy excised or irradiated with a high probability of cure)
* Malignant hepatic tumors
* Uncontrolled systemic infection
* Active viral infection with Human Immunodeficiency Virus (HIV) or Hepatitis type B or C
* Use of any experimental drug or therapy within 28 days prior to Day 1

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 488 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2014-01-22 (Actual); Study Completion 2016-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: C L Beach, PharmD, Study Director — Celgene Corporation
Locations (112):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - MD Anderson Cancer Center, Houston, Texas
- Australia (6):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Western Hospital, Footscray, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - St Vincent's Hospital, Fitzroy
- Austria (3):
  - Klinikum Wels-Grieskirchen GmbH, Wels, Upper Austria
  - Wilhelminenspital, I Medizinische Abt., Vienna, Vienna
  - Landeskliniken Salzburg Saint Johanns-Spital, III Medizinische Abteilung, Salzburg
- Belgium (5):
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir, Namur
  - Universitair Ziekenhuis Gent, Ghent, Oost-vlaanderen
  - Algemeen Ziekenhuis Sint-Jan, Bruges, West-vlaanderen
  - Centre Hospitalier de Jolimont-Lobbes, La Louvière
- Canada (10):
  - University of Alberta Hospital, Edmonton, Alberta
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Ottawa Hospital General Campus, Ottawa, Ontario
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Hospitalier de l'Université de Montréal pavilion Notre Dame, Montreal, Quebec
  - Hopital du Sacre Coeur de Montréal, Montreal, Quebec
  - Tom Baker Cancer Centre, Calgary
  - Princess Margaret Hospital, Ontario
- China (7):
  - The Third Hospital of Peking University, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peoples Hospital of Jiangsu Province, Jiangsu
  - Shanghai Ruijin Hospital, Shanghai
  - Shanghai Changhai Hospital,the Second Military Medical University, Shanghai
  - West China Hospital,Sichuan University, Sichuan
  - Tianjin Blood Disease Hospital, Tianjin
- Czechia (4):
  - Fakultni nemocnice Brno, Brno, Jihormoravsky Kraj
  - Fakultni nemocnice Olomouc, hemato-onkologicka klinika, Olomouc, Olomoucký kraj
  - Vseobecna Fakultni Nemocnice v Praze, Prague, Prague
  - Ustav hematologie a krevni transfuze, Prague, Prague
- France (13):
  - Centre Hospitalier Régional Universitaire, Hôpital de Hautepierre, Strasbourg, Alsace
  - Centre Hopitalier Universitaire Dupuytren, Limoges, Limousin Lorraine
  - Centre Hospitalier Universitaire de Toulouse, Toulouse, Midi-pyrénées
  - Centre Hospitalier Universitaire de Nice, Nice, Nice
  - CHRU d'Angers, Angers, Pays de la Loire Region
  - Centre Hospitalier Universitaire Nantes, Hotel Dieu, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire d'Amiens, Groupe Hospitalier Sud, Amiens, Picardie
  - Hôpital de la Conception, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de la Cote Basque, Aquitaine
  - Centre Hospitalier Universitaire de Lyon-Hôpital Edouard Herriot, Lyon
  - Hospital Avicenne, Service d'hematologie Clinique, Bobigny, Île-de-France Region
  - Hopital Percy Clamart, Clamart, Île-de-France Region
  - Hôpital Saint Louis, Paris, Île-de-France Region
- Germany (7):
  - Universitatsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - University of Rostock, Div. of Haematology and Oncology, Rostock, Mecklenburg-Vorpommern
  - Universitatsklinikum Essen, Zentrum fur Tumorforschung und Tumortherapie, Essen, Nordrhein-Westfallen
  - Heinrich-Heine-Universität Düsseldorf, Düesseldorf, North Rhine-Westphalia
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Jena, Jena, Thuringia
- Israel (7):
  - Soroka Medical Center, Beersheba, Beersheva
  - Assaf Harofeh Medical Centre, Beer Yaakov
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center - Tel Hashomer, Heart Institute, Tel Litwinsky
- Italy (12):
  - IRCCS Centro di Riferimento Oncologico di Basilicata di Rionero in Vulture, Rionero in Vulture, Potenza
  - Azienda Sanitaria Ospedaliera "San Luigi Gonzaga", Orbassano, Turin
  - Azienda Ospedaliera SS. Antonio E. Biagio E. Cesare Arrigo di Alessandria, Alessandria
  - Azienda Ospedaliera Universitaria - Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliera Policlinico di Bari, Bari
  - Azienda Ospedaliera Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli, Reggio Calabria
  - Azienda Policlinico Umberto I di Roma, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliero Universitaria S. Maria della Misericordia di Udine, Udine
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Universitair Medisch Centrum Groningen, Groningen, Netherlands
- Poland (5):
  - Katedra i Klinika Hematologii, Nowotworów Krwi i Transplantacji Szpiku, Wroclaw, Lower Silesian Voivodeship
  - Dolnoslaskie Centrum Transplantacji Komórkowych z Krajowym Bankiem Dawców Szpiku, Wroclaw, Lower Silesian Voivodeship
  - Instytut Hematologii i Transfuzjologii, Warsaw, Masovian Voivodeship
  - Samodzielny Publiczny SK im. A. Mieleckiego Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice, Silesian Voivodeship
  - Wojewodzki Szpital Specjalistczny im. Mikolaja Kopernika, Lódz, Łódź Voivodeship
- Russia (5):
  - City Clinical Hospital n.a. S. P. Botkin, Moscow
  - State Healthcare Institution "Nizhny Novgorod N.A. Semashko Regional Clinical Hospital", Nizhny Novgorod
  - Saint Petersburg State Academician I.P. Pavlov Medical University, Saint Petersburg
  - Saratov State Medical University, Saratov
  - Central City Hospital # 7, Yekaterinburg
- South Korea (7):
  - Samsung Medical Center, Gangnam-gu, Seoul
  - Seoul National University Hospital, Jongno-gu, Seoul
  - Yonsei University Health System, Seodaemun-gu, Seoul
  - Kyungpook National University Hospital, Daegu
  - Seoul Saint Mary's Hospital Seocho-gu, Seoul
  - Asan Medical Center, Seoul
  - Korea University Hospital at Guro, Seoul
- Spain (8):
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario La Fe, Valencia
- Taiwan (3):
  - Chang Gung Memorial Hospital, Kaohsiung, Niao-Sung Hsiang, Kaohsiung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital Pei-Tou District, Taipei
- United Kingdom (7):
  - Royal Marsden Hospital, Sutton, Surrey
  - Royal Bournemouth Hospital, Bournemouth
  - Barts and the London NHS Trust, London
  - King's College Hospital, London
  - Manchester Royal Infirmary, Manchester
  - Churchill Hospital, Oxford
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Seymour JF, Dohner H, Butrym A, Wierzbowska A, Selleslag D, Jang JH, Kumar R, Cavenagh J, Schuh AC, Candoni A, Recher C, Sandhu I, Del Castillo TB, Al-Ali HK, Falantes J, Stone RM, Minden MD, Weaver J, Songer S, Beach CL, Dombret H. Azacitidine improves clinical outcomes in older patients with acute myeloid leukaemia with myelodysplasia-related changes compared with conventional care regimens. BMC Cancer. 2017 Dec 14;17(1):852. doi: 10.1186/s12885-017-3803-6. PMID 29241450
- [Derived] Dombret H, Seymour JF, Butrym A, Wierzbowska A, Selleslag D, Jang JH, Kumar R, Cavenagh J, Schuh AC, Candoni A, Recher C, Sandhu I, Bernal del Castillo T, Al-Ali HK, Martinelli G, Falantes J, Noppeney R, Stone RM, Minden MD, McIntyre H, Songer S, Lucy LM, Beach CL, Dohner H. International phase 3 study of azacitidine vs conventional care regimens in older patients with newly diagnosed AML with >30% blasts. Blood. 2015 Jul 16;126(3):291-9. doi: 10.1182/blood-2015-01-621664. Epub 2015 May 18. PMID 25987659

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, international Phase 3 study conducted at 107 investigational sites in 18 countries including South Korea, China, Taiwan, Australia, Canada, United States, Poland, Russia, Czech Republic, Israel, France, Italy, Spain, Germany, United Kingdom, Belgium, Austria and the Netherlands.
Groups:
- Azacitidine (AZA): Azacitidine 75 mg/m2/day by subcutaneous injection [SC] for 7 days every 28 days, with a 21 day rest period (optimally for at least 6 cycles) plus best supportive care as needed, including antibiotics and blood product transfusions, growth factors, per physician's discretion.
- Conventional Care Regimens (CCR): CCRs included:
  * 1 Intensive Chemotherapy: Cytarabine 100-200 mg/m2 as a continuous intravenous infusion (CIVI) for 7 days and daunorubicin 45 to 60 mg/m² daily (QD) IV on Days 1, 2 and 3 or Idarubicin 9-12 mg/m² IV QD for 3 days. Consolidation Therapy (Cycle 2 and 3) = Cytarabine 100-200 mg/m2 as a CIVI for 3 to 7 days and daunorubicin 45 to 60 mg/m² QD or Idarubicin 9-12 mg/m² IV QD on Days 1 and 2. The first consolidation therapy started between Day 28 and Day 70 from start of induction therapy, upon recovery of absolute neutrophil count (ANC) above 1.0 x 10^9/L and platelets above 75 x 10^9/L. The second cycle started between Day 28 and Day 70 from start of first consolidation therapy. Best supportive care (BSC) of antibiotics and transfusions, were given as needed
  * 2 Low-dose cytarabine 20 mg subcutaneously twice a day (BID) for 10 days every 28 days, plus BSC
  * 3 BSC only = transfusion of blood products, antibiotics, antifungals and nutritional help
Period: Treatment Phase
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Started | 241 | 247
Treated Population | 236 (5 patients not treated with any drug regimen) | 240 (7 patients not treated with any drug regimen)
Safety Population | 236 (Received at least one dose of study medication and had at least 1 post dose safety assessment) | 235 (Received at least one dose of study medication and had at least 1 post dose safety assessment)
Evaluable Population | 179 (Did not meet criteria for exclusion, received ≥1 cycle of treatment and had ≥ 1 efficacy assessment) | 191 (Did not meet criteria for exclusion, received ≥1 cycle of treatment and had ≥ 1 efficacy assessment)
Completed | 24 (Participants who were continuing study treatment at the time of study closure) | 13 (Participants who were continuing study treatment at the time of study closure)
Not Completed | 217 | 234
Not completed — Adverse Event | 89 | 66
Not completed — Disease Progression | 16 | 21
Not completed — Withdrawal by Subject | 27 | 48
Not completed — Death | 53 | 58
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Miscellaneous | 32 | 39
Period: Survival Follow-Up Phase
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Started | 140 | 163
Completed | 16 | 27
Not Completed | 124 | 136
Not completed — Withdrawal by Subject | 5 | 8
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 116 | 124
Not completed — Alive at study closure | 1 | 3
Period: Extension Phase
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Started | 22 (2 participants did not enroll in the extension period.) | 0
Safety Population | 22 (Participants who enrolled in the extension phase) | 0
Completed | 0 | 0
Not Completed | 22 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Disease Progression | 9 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 5 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population is defined as all participants who were randomized, independent of whether they received study treatment or not.
Groups:
- Conventional Care Regimens (CCR): #1 Intensive Chemotherapy: Cytarabine 100-200 mg/m^2 as a continuous intravenous infusion (CIVI) for 7 days and daunorubicin 45 to 60 mg/m^² daily (QD) IV on Days 1, 2 and 3 or Idarubicin 9-12 mg/m^² IV QD for 3 days. Consolidation Therapy (Cycle 2 and 3) = Cytarabine 100-200 mg/m^2 as a CIVI for 3 to 7 days and daunorubicin 45 to 60 mg/m^² QD or Idarubicin 9-12 mg/m^² IV QD on Days 1 and 2. Consolidation therapy started between Day 28 and Day 70 from start of induction therapy, upon recovery of absolute neutrophil count (ANC) above 1.0 x 10^9/L and platelets above 75 x 10^9/L. The second cycle started between Day 28 and Day 70 from start of first consolidation therapy. Best supportive care (BSC) of antibiotics and transfusions, were given as needed. # 2 Low-dose cytarabine 20 mg SC twice a day (BID) for 10 days every 28 days, plus BSC # 3 BSC only includes transfusion of blood products, antibiotics, antifungals and nutritional help.
- Total: Total of all reporting groups
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR) | Total
Number analyzed (Participants) | 241 | 247 | 488
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (5.60) | 75.1 (5.57) | 75.2 (5.58)
Age, Customized [Number; unit: participants]
  <75 years | 103 | 120 | 223
  ≥75 years | 138 | 127 | 265
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 98 | 200
  Male | 139 | 149 | 288
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG performance status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity), 1 = Restricted activity but ambulatory, 2 = Ambulatory but unable to carry out work activities, 3 = Limited Self Care; 4 = Completely Disabled, No self care (Least Favorable Activity)
  participants
    0 = Fully Active | 54 | 57 | 111
    1 = Restrictive but Ambulatory | 132 | 132 | 264
    2 = Ambulatory but unable to work | 55 | 58 | 113
    3 = Limited Self Care | 0 | 0 | 0
    4 = Completely disabled | 0 | 0 | 0
World Health Organization Acute Myeloid Leukemia (AML) Classification [Number; unit: participants] — WHO categories include:
  1. Those with AML with recurrent genetic abnormalities. Includes subtypes with multiple chromosome translocations and mutations.
  2. Those with AML with myelodysplasia-related changes. Includes those with prior myelodysplastic syndrome (MDS) or myeloproliferative disease and has transformed to AML.
  3. Those with therapy related myeloid neoplasms and have had prior chemotherapy and/or radiation and subsequently develop AML or MDS
  4. Those with AML not otherwise specified and include subtypes that do not fall into the above categories.
  participants
    AML with myelodysplasia-related changes | 75 | 83 | 158
    Therapy-related myeloid neoplasms | 8 | 12 | 158
    AML with recurrent genetic abnormalities | 5 | 9 | 14
    AML not otherwise specified | 153 | 143 | 296
Bone Marrow-Blasts Counts [Mean (Standard Deviation); unit: Percentage of Bone Marrow Blasts] — Baseline clinical characteristics, including percentage of bone marrow blasts were assessed centrally and locally. Central values are included here. Baseline blasts were the last non-missing value on or prior to the date of randomization. The bone marrow blasts cells are not typically found in the circulating blood of healthy individuals. Abnormal immature white blood cells (blasts) fill the bone marrow and spill into the bloodstream.
  Percentage of Bone Marrow Blasts | 66.6 (24.71) | 70.2 (22.28) | 68.5 (23.56)

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimates for Overall Survival
Description: Overall Survival was defined as the time from randomization to death from any cause. Overall survival was calculated by the formula: date of death - date of randomization + 1. Participants surviving at the end of the follow-up period or who withdrew consent to follow-up were censored at the date of last contact. Participants who were lost to follow-up were censored at the date last known alive.
Time Frame: Day 1 (randomization) to 40 months
Population: The intent-to-treat (ITT) population was defined as all participants who were randomized, independent of whether they received study treatment or not. Includes participants who died and participants who were censored
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Conventional Care Regimens (CCR): CCRs included: #1 Intensive Chemotherapy: Cytarabine 100-200 mg/m^2 as a continuous intravenous infusion (CIVI) for 7 days and daunorubicin 45 to 60 mg/m^² daily (QD) IV on Days 1, 2 and 3 or Idarubicin 9-12 mg/m^² IV QD for 3 days. Consolidation Therapy (Cycle 2 and 3) = Cytarabine 100-200 mg/m^2 as a CIVI for 3 to 7 days and daunorubicin 45 to 60 mg/m^² QD or Idarubicin 9-12 mg/m^² IV QD on Days 1 and 2. The first consolidation therapy started between Day 28 and Day 70 from start of induction therapy, upon recovery of absolute neutrophil count (ANC) above 1.0 x 10^9/L and platelets above 75 x 10^9/L. The second cycle started between Day 28 and Day 70 from start of first consolidation therapy. Best supportive care (BSC) of antibiotics and transfusions, were given as needed # 2 Low-dose cytarabine 20 mg subcutaneously twice a day (BID) for 10 days every 28 days, plus BSC # 3 BSC only = transfusion of blood products, antibiotics, antifungals and nutritional help
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Number analyzed (Participants) | 241 | 247
months | 10.4 [8.0 to 12.7] | 6.5 [5.0 to 8.6]
Statistical Analysis 1: Comparison: Azacitidine (AZA) vs Conventional Care Regimens (CCR); Test type: Superiority or Other; p = 0.0829, Log Rank; The p-value is two-sided from an unstratified log-rank test; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.69 to 1.02] — The hazard ratio is from a Cox proportional hazards model stratified by ECOG performance status and cytogenetic risk status
Statistical Analysis 2: Comparison: Azacitidine (AZA) vs Conventional Care Regimens (CCR); Test type: Superiority; p = 0.1009, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.69 to 1.03] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: One-year Overall Survival Rate
Description: Kaplan Meier methods were used to estimate the 1-year survival probabilities for time to death from any cause. Estimates of the 1-year (365 day) survival probabilities and corresponding 95% confidence intervals (CI) were presented by treatment group. The CI for the difference in the 1-year survival probabilities was derived using Greenwoods variance estimate.
Time Frame: From Day 1 (randomization) to 40 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Conventional Care Regimen: CCRs included: #1 Intensive Chemotherapy: Cytarabine 100-200 mg/m^2 as a continuous intravenous infusion (CIVI) for 7 days and daunorubicin 45 to 60 mg/m^² daily (QD) IV on Days 1, 2 and 3 or Idarubicin 9-12 mg/m^² IV QD for 3 days. Consolidation Therapy (Cycle 2 and 3) = Cytarabine 100-200 mg/m^2 as a CIVI for 3 to 7 days and daunorubicin 45 to 60 mg/m^² QD or Idarubicin 9-12 mg/m^² IV QD on Days 1 and 2. The first consolidation therapy started between Day 28 and Day 70 from start of induction therapy, upon recovery of absolute neutrophil count (ANC) above 1.0 x 10^9/L and platelets above 75 x 10^9/L. The second cycle started between Day 28 and Day 70 from start of first consolidation therapy. Best supportive care (BSC) of antibiotics and transfusions, were given as needed # 2 Low-dose cytarabine 20 mg subcutaneously twice a day (BID) for 10 days every 28 days, plus BSC # 3 BSC only = transfusion of blood products, antibiotics, antifungals and nutritional help
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 241 | 247
percentage of participants | 46.5 [40.1 to 52.7] | 34.3 [28.3 to 40.3]
Statistical Analysis 1: Comparison: Azacitidine (AZA) vs Conventional Care Regimen; Test type: Superiority or Other; Difference = 12.26, 95% CI 2-sided [3.5 to 21.0] — Estimates of the 1-year (365 day) survival probabilities and corresponding 95% confidence intervals (CI) were presented by treatment group. The CI for the difference in the 1-year survival probabilities was derived using Greenwoods variance estimate

3. Secondary Outcome: Event-free Survival (EFS)
Description: Event-free survival was defined as the interval from the date of randomization to the date of treatment failure, progressive disease, relapse after complete remission (CR) or complete remission with incomplete blood count recovery (CRi), death from any cause, or lost to follow-up, whichever occurs first. Participants who were still alive without any of these events were censored at the date of their last response assessment.
Time Frame: Day 1 (randomization) to date of treatment failure, progressive disease, relapse after Complete Remission (CR) or Complete remission with incomplete blood count recovery (CRi), death from any cause. Day 1 (randomization) to 40 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Number analyzed (Participants) | 241 | 247
months | 6.7 [5.0 to 8.8] | 4.8 [3.8 to 6.0]
Statistical Analysis 1: Comparison: Azacitidine (AZA) vs Conventional Care Regimens (CCR); Median is estimated from a Kaplan-Meier distribution of EFS; Test type: Superiority or Other; p = 0.1495, Log Rank; 2 sided unstratified; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.72 to 1.05] — The hazard ratio is from an unstratified Cox proportional hazards model

4. Secondary Outcome: Relapse-Free Survival (RFS) for Participants Who Achieved a Complete Remission (CR) or Complete Remission With Incomplete Blood Count Recovery (CRi)
Description: Relapse-free survival was defined as the interval from the date of first documented CR or CRi to the date of relapse, death from any cause, or lost to follow-up, whichever occurred first. Participants who were still alive and in continuous CR or CRi were censored at the date of their last response assessment.
Time Frame: Day 1 of first documented CR or CRi to the date of relapse, death from any cause, or lost to follow-up. Day 1 (randomization) to 40 months
Population: Participants who achieved a CR or CRi
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 67 | 62
months | 9.3 [6.7 to 12.4] | 10.5 [7.3 to 12.3]
Statistical Analysis 1: Comparison: Azacitidine (AZA) vs Conventional Care Regimen; Median is estimated from a Kaplan-Meier distribution of RFS; Test type: Superiority or Other; p = 0.5832, Log Rank; 2 sided unstratified; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.75 to 1.66] — The hazard ratio is from an unstratified Cox proportional hazards model

5. Secondary Outcome: Percentage of Participants Who Achieved a Morphologic CR + CRi as Determined by the Independent Review Committee (IRC) Based on International Working Group (IWG) Response Criteria for Acute Myeloid Leukemia (AML)
Description: A complete remission (CR) is defined as a leukemia-free state defined as less than 5% blasts in a BM aspirate with marrow spicules and with at least 200 nucleated cells (there should be no blasts with Auer rods), an absolute neutrophil count (ANC) of ≥ 1 x 10^9/L, a platelet count ≥ 100 x 10^9/L, and transfusion independence (no transfusions for 1 week prior to each assessment). No duration of these findings is required for confirmation of this response. A CR with incomplete blood count recovery (CRi) is defined as <5% BM blasts with the ANC count < 1 x 10^9/L and/or the platelet count may be < 100 x 10^9/L. Where the date of the hematology assessment used is the earliest on or following the date of the BM sample up to 8 days after the BM date.
Time Frame: Day 1 (randomization) to 40 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Number analyzed (Participants) | 241 | 247
percentage of participants | 27.8 | 25.1
Statistical Analysis 1: Comparison: Azacitidine (AZA) vs Conventional Care Regimens (CCR); Test type: Superiority or Other; p = 0.5384, Fisher Exact; P-value is from Fishers exact test

6. Secondary Outcome: Duration of Remission Assessed by the IRC Based on Kaplan-Meier Estimates
Description: The time from the date CR or CRi was first documented until the date of documented relapse from CR/CRi. Duration of remission was defined only for those participants who achieved a CR or CRi, as determined by the IRC. Participants who were lost to follow-up without documented relapse, or were alive at last follow-up without documented relapse were censored at the date of their last response assessment.
Time Frame: Day 1 (randomization) to 40 months; date of the first documented CR or CRi until date of first documented relapse.
Population: Includes those who achieved a CR or CRi and assessed by the IRC; numbers of ITT participants in each treatment group
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 67 | 62
months | 10.4 [7.2 to 15.2] | 12.3 [9.0 to 17.0]

7. Secondary Outcome: Number of Participants Who Achieved a Cytogenetic Complete Response (CRc-10) as Determined by the IRC.
Description: The CRc is a normal karyotype defined as no clonal abnormalities after review of at least 10 metaphases using conventional cytogenetic techniques. Cytogenetic complete remission rate (CRc) is when the following criteria are met: 1) CR criteria met and 2) an abnormal karyotype is present at baseline and 3) there is reversion to normal karyotype at the time of CR (based on ≥ 10 metaphases), where date of cytogenetic sample = date of BM sample used for the CR assessment
Time Frame: Day 1 (randomization) to 40 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Number analyzed (Participants) | 241 | 247
participants | 5 | 15
Statistical Analysis 1: Comparison: Azacitidine (AZA) vs Conventional Care Regimens (CCR); Test type: Superiority or Other; p = 0.0376, Fisher Exact; P-value is from Fishers exact test

8. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AEs = any noxious, unintended, or untoward medical occurrence that may appear or worsen during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, regardless of cause. Serious AE (SAE) = any AE which results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; constitutes an important medical event. The severity of AEs were graded based upon the participants symptoms according to the Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0); AEs were evaluated for severity according to the following scale: Grade 1 = Mild - transient or mild discomfort; no medical intervention required; Grade 2 = Moderate - mild to moderate limitation in activity; Grade 3 = Severe; Grade 4 = Life threatening; Grade 5 = Death
Time Frame: Day 1 (randomization) up to last visit completed; final data cut off of 28 Feb 2017
Population: Safety population = all randomized participants who received at least 1 dose of study drug and had 1 post-dose safety assessment. Because the BSC only regimen consisted of blood products or antibiotics given as needed, those assigned to BSC only were included in the safety population if they had at least 1 post-randomization safety assessment.
Measure: Number; unit: participants
Groups:
- Conventional Care Regimen #3 Best Supportive Care Only: Best supportive care included red blood cell (RBC) or whole blood transfusions, fresh frozen plasma transfusions, platelet transfusions, antibiotic and/or antifungal therapy, and nutritional support.
- Conventional Care Regimen #2 Low-dose Cytarabine: Low-dose cytarabine 20 mg SC injection twice a day (BID) for 10 days, every 28 days (optimally for at least 4 cycles) until the end of the study, unless participants were discontinued from the treatment. Best supportive care as needed, including antibiotics and transfusions, per physicians discretion.
- Conventional Care Regimen #1 Intensive Chemotherapy: Induction Therapy included Cytarabine 100-200 mg/m^2 as a continuous intravenous infusion (IV) for 7 days plus daunorubicin 45 to 60 mg/m^² daily IV on Days 1, 2 and 3 or Idarubicin 9-12 mg/m^² IV daily for 3 days as an alternative to daunorubicin (Cycle 1). Consolidation Therapy (Cycle 2 and 3) Cytarabine 100-200 mg/m^2 as a continuous IV infusion for a total of 3 to 7 days plus daunorubicin 45 to 60 mg/m^² daily or Idarubicin 9-12 mg/m^² IV daily on Days 1 and 2. The first consolidation therapy started between Day 28 and Day 70 from commencement of induction therapy, upon recovery of absolute neutrophil count (ANC) to at least 1.0 x 10^9/L and platelets to at least 75 x 10^9/L. The second consolidation cycle, if given, started between Day 28 and Day 70 from commencement of the first consolidation therapy. Participants could receive BSC as needed, including antibiotics and transfusions, physicians discretion.
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen #3 Best Supportive Care Only | Conventional Care Regimen #2 Low-dose Cytarabine | Conventional Care Regimen #1 Intensive Chemotherapy
Number analyzed (Participants) | 236 | 40 | 153 | 42
participants
  At least one Treatment Emergent AE | 234 | 36 | 153 | 42
  At least one TEAE related to study drug | 188 | 0 | 124 | 39
  Grade 3-4 adverse event | 207 | 26 | 141 | 37
  Grade 3-4 adverse event related to any study drug | 125 | 0 | 90 | 29
  At least one Grade 5 (leading to death) TEAE | 56 | 23 | 38 | 9
  Grade 5 adverse event related to any study drug | 12 | 0 | 10 | 4
  Serious TEAE | 188 | 30 | 118 | 27
  Serious TEAE related to any study drug | 87 | 0 | 56 | 14
  TEAE leading to discontinuation of study drug | 110 | 0 | 68 | 11
  Study drug-related TEAE leading to discontinuation | 22 | 0 | 20 | 5
  TEAE leading to study drug dose reduction | 8 | 0 | 2 | 2
  TEAE leading to study drug dose interruption | 116 | 0 | 61 | 4
  TEAE causing study drug dose reduction/disruption | 13 | 0 | 7 | 0

9. Secondary Outcome: Health Related Quality of Life (HRQoL): Change From Baseline in the European Organization for Research and Treatment of Cancer Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Fatigue Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Fatigue Scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate reduction in fatigue (i.e. improvement in symptom) and positive values indicate increases in fatigue (i.e. worsening of symptom).
Time Frame: Baseline to Cycle 3; at approximately 3 months
Population: The HRQoL Evaluable population included only participants with a baseline QoL assessment and at least 1 follow-up assessment. Time windows were applied post-hoc to increase the size of the analyzable population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Number analyzed (Participants) | 135 | 101
units on a scale | -1.5 (24.69) | -1.9 (27.54)

10. Secondary Outcome: Health Related Quality of Life (HRQoL): Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Fatigue Domain
Description: as for outcome 9
Time Frame: Baseline to Cycle 5, at approximately 5 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Number analyzed (Participants) | 112 | 66
units on a scale | -2.8 (27.36) | -7.1 (27.61)

11. Secondary Outcome: Health Related Quality of Life (HRQoL): Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Fatigue Domain
Description: as for outcome 9
Time Frame: Baseline to Cycle 7, at approximately 7 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Number analyzed (Participants) | 94 | 53
units on a scale | -6.1 (26.90) | -12.2 (30.45)

12. Secondary Outcome: Health Related Quality of Life (HRQoL): Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Fatigue Domain
Description: as for outcome 9
Time Frame: Baseline to Cycle 9, at approximately 9 months
Population: The HRQoL Evaluable population included only participants with a baseline QoL assessment and at least 1 follow-up assessment. Time windows were applied post-hoc to increase the size of the analyzable population. .
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Number analyzed (Participants) | 80 | 36
units on a scale | -9.0 (27.90) | -10.2 (33.85)

13. Secondary Outcome: Health Related Quality of Life (HRQoL): Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Fatigue Domain
Description: as for outcome 9
Time Frame: Baseline to End of Study; at approximately 11-12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Number analyzed (Participants) | 87 | 80
units on a scale | 8.9 (33.54) | 6.1 (34.19)

14. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Dyspnea
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Dyspnea scale is scored between 0 and 100, with a high score indicating a higher level of symptoms. Negative change from Baseline values indicate decreased dyspnea (i.e. improvement in symptom) and positive values indicate increased dyspnea (i.e. worsening of symptom).
Time Frame: Baseline to Cycle 3, at approximately 3 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 136 | 101
units on a scale | 5.1 (26.88) | -1.7 (30.69)

15. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Dyspnea
Description: as for outcome 14
Time Frame: Baseline to Cycle 5, at approximately 5 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 112 | 66
units on a scale | 3.9 (27.49) | -6.6 (28.18)

16. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Dyspnea
Description: as for outcome 14
Time Frame: Baseline to Cycle 7, at approximately 7 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 94 | 53
units on a scale | 0.4 (29.93) | -8.8 (28.61)

17. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Dyspnea
Description: as for outcome 14
Time Frame: Baseline to Cycle 9, at approximately 9 months
Population: The HRQoL Evaluable population included only participants with a baseline QoL assessment and at least 1 follow-up assessment. Time windows were applied post-hoc to increase the size of the analyzable population. The analysis included 157 from the azacitidine group and 134 in the CCR group, a smaller number than the ITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 81 | 36
units on a scale | -4.9 (26.93) | -2.8 (26.87)

18. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Dyspnea
Description: as for outcome 14
Time Frame: Baseline to end of study, at approximately 11-12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 87 | 80
units on a scale | 12.6 (31.43) | 6.3 (35.22)

19. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Physical Functioning Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 PhysicalFunctioning Scale is scored between 0 and 100, with a high score indicating better functioning. Negative change from Baseline values indicate deterioration in functioning and positive values indicate improvement.
Time Frame: Baseline to Cycle 3, at approximately 3 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 136 | 102
units on a scale | -4.2 (17.98) | -0.3 (18.85)

20. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Physical Functioning Domain
Description: as for outcome 19
Time Frame: Baseline to Cycle 5, at approximately 5 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 112 | 67
units on a scale | -4.4 (19.25) | -1.3 (20.41)

21. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Physical Functioning Domain
Description: as for outcome 19
Time Frame: Baseline to Cycle 7, at approximately 7 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 94 | 54
units on a scale | 1.6 (18.75) | 1.5 (23.08)

22. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Physical Functioning Domain
Description: as for outcome 19
Time Frame: Baseline to Cycle 9, at approximately 9 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 81 | 36
units on a scale | 3.5 (18.26) | -0.4 (22.81)

23. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Physical Functioning Domain
Description: as for outcome 19
Time Frame: Baseline to end of study, at approximately 11-12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 87 | 81
units on a scale | -13.0 (26.74) | -9.4 (26.43)

24. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Global Health Status-/Quality of Life Domain
Description: The European Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life (QOL) questionnaire (EORTC QLQ-C30) is a 30-question tool used to assess the overall quality of life in cancer patients. It consists of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, Role, Cognitive, Emotional, Social), and 9 symptom scales/items (Fatigue, Nausea and Vomiting, Pain, Dyspnea, Sleep Disturbance, Appetite Loss, Constipation, Diarrhea, Financial Impact). The EORTC QLQ-C30 Global Health Status/QOL scale is scored between 0 and 100, with a high score indicating better Global Health Status/QOL. Negative change from Baseline values indicate deterioration in Global Health Status/QOL and positive values indicate improvement.
Time Frame: Baseline to Cycle 3, at approximately 3 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 134 | 101
units on a scale | 0.9 (20.97) | 3.8 (26.42)

25. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Global Health Status-/Quality of Life Domain
Description: as for outcome 24
Time Frame: Baseline to Cycle 5, at approximately 5 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 112 | 66
units on a scale | 1.6 (22.50) | 9.0 (24.82)

26. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Global Health Status-/Quality of Life Domain
Description: as for outcome 24
Time Frame: Baseline to Cycle 7, at approximately 7 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 94 | 52
units on a scale | 5.1 (25.84) | 8.7 (27.91)

27. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Global Health Status-/Quality of Life Domain
Description: as for outcome 24
Time Frame: Baseline to Cycle 9, at approximately 9 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 80 | 36
units on a scale | 7.8 (27.28) | 10.4 (23.09)

28. Secondary Outcome: HRQoL: Change From Baseline in the EORTC QLQ-C30 Global Health Status-/Quality of Life Domain
Description: as for outcome 24
Time Frame: Baseline to end of study, at approximately 11-12 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 87 | 80
units on a scale | -4.4 (29.20) | -6.1 (27.90)

29. Secondary Outcome: Healthcare Resource Utilization (HRU): Number of Inpatient Hospitalizations
Description: HRU was defined as any consumption of healthcare resources directly or indirectly related to the treatment of the patient. HRU Analysis may help in evaluating potential costs and budget impact of new treatments from a payer perspective.
Time Frame: Day 1 (randomization) to 40 months
Population: HRU was analyzed for the HRQoL Evaluable Population, a smaller sample than either the ITT population or safety population. Duration of therapy differed between treatment groups. Rate-per-patient year values adjust for these differences.
Measure: Number; unit: participants
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Number analyzed (Participants) | 157 | 134
participants | 139 | 111

30. Secondary Outcome: Healthcare Resource Utilization (HRU): Rate of Inpatient Hospitalizations Per Year
Description: HRU was defined as any consumption of healthcare resources directly or indirectly related to the treatment of the patient. HRU Analysis may help in evaluating potential costs and budget impact of new treatments from a payer perspective. The rate of inpatient hospitalizations per patient year was calculated as the total number of hospitalizations divided by the total number of patient-years followed in the study period. Patient-years (PY) were calculated as the duration from baseline to last available HRQL assessment for each patient.
Time Frame: Day 1 (randomization) to 40 months
Population: as for outcome 29
Measure: Number; unit: hospitalizations per patient year
Arm/Group | Azacitidine (AZA) | Conventional Care Regimens (CCR)
Number analyzed (Participants) | 157 | 134
hospitalizations per patient year | 7.95 | 4.82

31. Secondary Outcome: HRU: Number of Participants Receiving Transfusions
Description: Count of study participants who had transfusions during the treatment phase. HRU is defined as any consumption of healthcare resources directly or indirectly related to the treatment of the patient. HRU Analysis may help in evaluating potential costs and budget impact of new treatments from a payer perspective.
Time Frame: Day 1 (randomization) to 40 months
Population: as for outcome 29
Measure: Number; unit: participants
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 157 | 134
participants | 154 | 134
Statistical Analysis 1: Comparison: Azacitidine (AZA) vs Conventional Care Regimen; Test type: Superiority or Other; p = 0.0721, negative binomial regression analysis; Relative Ratio = 0.79, 95% CI 2-sided [0.62 to 1.02]

32. Secondary Outcome: HRU: Rate of Transfusions Per Patient Year
Description: HRU is defined as any consumption of healthcare resources directly or indirectly related to the treatment of the patient. HRU Analysis may help in evaluating potential costs and budget impact of new treatments from a payer perspective. The rate of transfusions per patient year was calculated as the total number of transfusions divided by the total number of patient-years followed in the study period. Patient-years (PY) were calculated as the duration from baseline to last available HRQL assessment for each patient.
Time Frame: Day 1 (randomization) to 40 months
Population: as for outcome 29
Measure: Number; unit: transfusions per patient year
Arm/Group | Azacitidine (AZA) | Conventional Care Regimen
Number analyzed (Participants) | 157 | 134
transfusions per patient year | 34.23 | 36.04

33. Secondary Outcome: Number of Participants in the Extension Phase With Treatment Emergent Adverse Events (TEAEs)
Description: as for outcome 8
Time Frame: From the date of informed consent for the Extension Phase through to the date of last dose of study drug + 28 days up to last visit completed 24 July 2016; maximum duration of exposure to Azacitidine was 871 days
Population: Safety population includes those enrolled in the extension phase who received at least one dose of study drug.
Measure: Number; unit: participants
Units Other Than Participants: participants
Arm/Group | Azacitidine (AZA)
Number analyzed (Participants) | 22
participants
  At least one Treatment Emergent AE | 20
  At least one TEAE related to study drug | 13
  At least one Grade 3-4 adverse event | 13
  At least 1 Grade 3-4 TEAE related to study drug | 7
  At least 1 Grade 5 TEAE | 4
  At least 1 Grade 5 TEAE related to study drug | 0
  At least 1 serious TEAE | 10
  At least 1 serious TEAE related to study drug | 1
  At least one serious Grade 3-4 TEAE | 8
  TEAE leading to discontinuation of study drug | 3
  Study drug-related TEAE leading to discontinuation | 1
  TEAE leading to study drug dose reduction | 1
  TEAE leading to study drug dose interruption only | 17
  TEAE causing study dose reduction/interruption | 2

ADVERSE EVENTS:
Time Frame: From first dose to 1) last dose + 28 days for azacitidine and low-dose cytarabine; 2) last dose + 70 days for intensive chemotherapy; 3) discontinuation for BSC only. Median duration was 191.5, 65.0, 125.0, 124.5 and 360.0 days for each group respectively
Description: 3) discontinuation for BSC only. Median duration was 191.5, 65.0, 125.0, 124.5 and 360.0 days for each group respectively.
  AEs reported for the Azacitidine group are those that occurred in the treatment phase, AEs reported in the Azacitidine extension group occurred during extension phase
Groups:
- Azacitidine; Azacitidine-extension: Azacitidine 75 mg/m^2/day by subcutaneous injection [SC] for 7 days every 28 days, with a 21 day rest period (optimally for at least 6 cycles) plus best supportive care as needed, including antibiotics and blood product transfusions, growth factors, per physician's discretion
- BSC Only: Transfusion of blood products, antibiotics, antifungals and nutritional help
- Low-dose Cytarabine: Low-dose cytarabine 20 mg subcutaneously twice a day (BID) for 10 days every 28 days, plus BSC
- Intensive Chemotherapy: Cytarabine 100-200 mg/m^2 as a continuous intravenous infusion (CIVI) for 7 days and daunorubicin 45 to 60 mg/m^² daily (QD) IV on Days 1, 2 and 3 or Idarubicin 9-12 mg/m^² IV QD for 3 days. Consolidation Therapy (Cycle 2 and 3) = Cytarabine 100-200 mg/m^2 as a CIVI for 3 to 7 days and daunorubicin 45 to 60 mg/m^² QD or Idarubicin 9-12 mg/m^² IV QD on Days 1 and 2. The first consolidation therapy started between Day 28 and Day 70 from start of induction therapy, upon recovery of absolute neutrophil count (ANC) above 1.0 x 10^9/L and platelets above 75 x 10^9/L. The second cycle started between Day 28 and Day 70 from start of first consolidation therapy. Best supportive care (BSC) of antibiotics and transfusions, were given as needed
Arm/Group | Azacitidine | BSC Only | Low-dose Cytarabine | Intensive Chemotherapy | Azacitidine-extension
Serious Adverse Events (participants affected / at risk) | 188/236 | 30/40 | 118/153 | 27/42 | 10/22
Other Adverse Events (participants affected / at risk) | 226/236 | 33/40 | 151/153 | 42/42 | 18/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=236) | BSC Only (N=40) | Low-dose Cytarabine (N=153) | Intensive Chemotherapy (N=42) | Azacitidine-extension (N=22)
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 10 | 1 | 11 | 0 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
FEBRILE BONE MARROW APLASIA (Blood and lymphatic system disorders) | 2 | 0 | 3 | 0 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 59 | 12 | 38 | 7 | 4
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 4 | 0 | 1 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 5 | 1 | 3 | 1 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 6 | 0 | 14 | 0 | 0
THROMBOTIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 2 | 0 | 1 | 0 | 0
ACUTE LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 3 | 0 | 0 | 1 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 7 | 1 | 3 | 2 | 0
CARDIAC ARREST (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 2 | 0 | 1 | 1 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 1 | 0 | 2 | 1 | 0
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
LEFT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0 | 1 | 0
PERICARDITIS (Cardiac disorders) | 1 | 0 | 1 | 0 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
CATARACT (Eye disorders) | 1 | 0 | 0 | 0 | 0
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 1 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
ANAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
ASCITES (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
COLITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 4 | 0 | 4 | 0 | 0
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
DUODENAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
ENTERITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1 | 4 | 0 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
ILEUS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
MELAENA (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
MOUTH HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
RECTAL ULCER (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
ASTHENIA (General disorders) | 4 | 1 | 3 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 2 | 1 | 0
CHILLS (General disorders) | 1 | 0 | 1 | 0 | 0
DEATH (General disorders) | 3 | 0 | 2 | 0 | 0
FATIGUE (General disorders) | 3 | 0 | 1 | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0 | 1 | 0 | 0
HYPERTHERMIA (General disorders) | 1 | 0 | 0 | 0 | 0
INJECTION SITE EXTRAVASATION (General disorders) | 1 | 0 | 0 | 0 | 0
INJECTION SITE REACTION (General disorders) | 2 | 0 | 0 | 0 | 0
MALAISE (General disorders) | 1 | 0 | 0 | 0 | 0
MULTI-ORGAN FAILURE (General disorders) | 1 | 0 | 2 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 0 | 0 | 0
PAIN (General disorders) | 1 | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 25 | 3 | 16 | 2 | 0
SUDDEN CARDIAC DEATH (General disorders) | 1 | 0 | 1 | 0 | 0
SUDDEN DEATH (General disorders) | 2 | 0 | 0 | 0 | 0
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 1 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
ANAPHYLACTIC SHOCK (Immune system disorders) | 1 | 0 | 0 | 0 | 0
ABSCESS NECK (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ABSCESS SOFT TISSUE (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ACUTE SINUSITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
AEROMONA INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
APPENDICITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ASPERGILLUS INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0
BACTERAEMIA (Infections and infestations) | 2 | 0 | 1 | 0 | 1
BRONCHITIS (Infections and infestations) | 3 | 0 | 1 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 4 | 1 | 1 | 0 | 0
BRONCHOPULMONARY ASPERGILLOSIS (Infections and infestations) | 3 | 1 | 0 | 0 | 1
CANDIDA INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 5 | 4 | 3 | 1 | 0
CELLULITIS ORBITAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 2 | 0 | 1 | 0 | 0
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 | 0 | 1 | 0 | 0
CORYNEBACTERIUM SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
CYSTITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
DEVICE RELATED SEPSIS (Infections and infestations) | 2 | 0 | 0 | 0 | 0
DIVERTICULITIS (Infections and infestations) | 4 | 0 | 0 | 0 | 0
ENTEROBACTER PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1 | 1 | 0 | 0
ENTEROCOCCAL SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
EPIGLOTTITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ESCHERICHIA BACTERAEMIA (Infections and infestations) | 3 | 0 | 1 | 0 | 0
ESCHERICHIA INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 4 | 0 | 0 | 0 | 0
FURUNCLE (Infections and infestations) | 1 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 1 | 0 | 0
GASTROENTERITIS CLOSTRIDIAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
GASTROINTESTINAL FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0
GROIN ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0 | 0 | 0 | 0
INFECTED CYST (Infections and infestations) | 1 | 0 | 0 | 0 | 0
INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 1
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 0 | 0 | 1 | 0 | 0
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0
KLEBSIELLA SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
LIVER ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 1
LOBAR PNEUMONIA (Infections and infestations) | 2 | 0 | 2 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1 | 1 | 0 | 0
LUNG ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
LUNG INFECTION (Infections and infestations) | 2 | 0 | 1 | 0 | 0
MUMPS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
NEUTROPENIC SEPSIS (Infections and infestations) | 7 | 2 | 4 | 1 | 0
ORAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
OROPHARYNGITIS FUNGAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PERIORBITAL CELLULITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0
PERIRECTAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PERITONITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
PHARYNGITIS (Infections and infestations) | 2 | 0 | 2 | 0 | 0
PHARYNGOTONSILLITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 48 | 3 | 29 | 3 | 2
PNEUMONIA FUNGAL (Infections and infestations) | 3 | 0 | 1 | 0 | 0
PNEUMONIA KLEBSIELLA (Infections and infestations) | 0 | 0 | 1 | 0 | 0
PNEUMONIA MYCOPLASMAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PNEUMONIA PARAINFLUENZAE VIRAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PNEUMONIA PSEUDOMONAS AERUGINOSA (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 | 0 | 1 | 0 | 0
PNEUMONIA STREPTOCOCCAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
PSEUDOMEMBRANOUS COLITIS (Infections and infestations) | 3 | 0 | 1 | 0 | 0
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 0 | 0 | 1 | 0 | 1
PSEUDOMONAL SEPSIS (Infections and infestations) | 3 | 0 | 2 | 0 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 2 | 2 | 0 | 0
SEPSIS (Infections and infestations) | 12 | 1 | 9 | 2 | 0
SEPTIC SHOCK (Infections and infestations) | 4 | 1 | 4 | 4 | 0
SINUSITIS (Infections and infestations) | 3 | 0 | 0 | 0 | 1
SINUSITIS FUNGAL (Infections and infestations) | 0 | 0 | 0 | 1 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 1 | 0 | 0 | 1 | 0
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
SYSTEMIC CANDIDA (Infections and infestations) | 0 | 0 | 0 | 0 | 1
TONSILLITIS (Infections and infestations) | 0 | 0 | 2 | 0 | 0
TOOTH INFECTION (Infections and infestations) | 2 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 7 | 1 | 3 | 0 | 0
UROSEPSIS (Infections and infestations) | 2 | 0 | 0 | 0 | 0
VAGINITIS GARDNERELLA (Infections and infestations) | 0 | 0 | 1 | 0 | 0
VULVAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0
ZYGOMYCOSIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
ALLERGIC TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
TRANSFUSION REACTION (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
TROPONIN INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0
URINE OUTPUT DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0
CACHEXIA (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 0 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
HAEMARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 | 12 | 17 | 0 | 1
CHLOROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0
LEUKAEMIC INFILTRATION BRAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
OVARIAN CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 2 | 0 | 1 | 0
CEREBRAL INFARCTION (Nervous system disorders) | 2 | 0 | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 2 | 0 | 0
COGNITIVE DISORDER (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
CONVULSION (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 5 | 0 | 0 | 0 | 1
FEBRILE CONVULSION (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 2 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
ORTHOSTATIC INTOLERANCE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 2 | 1 | 0 | 0 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 4 | 0 | 2 | 1 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
BLADDER MASS (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
HAEMATURIA (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
RENAL COLIC (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
RENAL FAILURE (Renal and urinary disorders) | 3 | 0 | 2 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3 | 0 | 2 | 1 | 0
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
RENAL TUBULAR NECROSIS (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 3 | 1 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
PULMONARY ALVEOLAR HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 6 | 2 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 2 | 1 | 0 | 0 | 0
HAEMATOMA (Vascular disorders) | 2 | 0 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0 | 0 | 0
HYPOTENSION (Vascular disorders) | 4 | 1 | 0 | 0 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0 | 0 | 0 | 0
PHLEBITIS (Vascular disorders) | 1 | 0 | 0 | 0 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azacitidine (N=236) | BSC Only (N=40) | Low-dose Cytarabine (N=153) | Intensive Chemotherapy (N=42) | Azacitidine-extension (N=22)
ANAEMIA (Blood and lymphatic system disorders) | 41 | 3 | 32 | 7 | 4
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 28 | 2 | 21 | 12 | 0
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 13 | 2 | 11 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 22 | 0 | 15 | 6 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 69 | 1 | 43 | 14 | 6
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 60 | 2 | 37 | 9 | 6
ATRIAL FIBRILLATION (Cardiac disorders) | 12 | 2 | 9 | 1 | 1
TACHYCARDIA (Cardiac disorders) | 5 | 3 | 2 | 2 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 | 4 | 4 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 30 | 3 | 16 | 7 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 19 | 0 | 6 | 6 | 0
CONSTIPATION (Gastrointestinal disorders) | 99 | 9 | 42 | 16 | 1
DIARRHOEA (Gastrointestinal disorders) | 87 | 5 | 34 | 21 | 5
DYSPEPSIA (Gastrointestinal disorders) | 16 | 2 | 14 | 6 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 14 | 1 | 7 | 4 | 3
MOUTH ULCERATION (Gastrointestinal disorders) | 11 | 1 | 8 | 1 | 0
NAUSEA (Gastrointestinal disorders) | 93 | 3 | 43 | 24 | 3
STOMATITIS (Gastrointestinal disorders) | 20 | 2 | 14 | 4 | 2
VOMITING (Gastrointestinal disorders) | 53 | 3 | 24 | 8 | 3
ASTHENIA (General disorders) | 53 | 8 | 32 | 5 | 6
CATHETER SITE PAIN (General disorders) | 3 | 0 | 1 | 3 | 0
CHILLS (General disorders) | 11 | 1 | 7 | 4 | 0
FATIGUE (General disorders) | 53 | 10 | 19 | 4 | 3
INJECTION SITE ERYTHEMA (General disorders) | 29 | 0 | 0 | 0 | 1
INJECTION SITE PAIN (General disorders) | 12 | 0 | 1 | 0 | 1
INJECTION SITE REACTION (General disorders) | 30 | 0 | 0 | 0 | 0
MALAISE (General disorders) | 7 | 2 | 3 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 8 | 0 | 14 | 3 | 0
OEDEMA (General disorders) | 8 | 0 | 3 | 1 | 2
OEDEMA PERIPHERAL (General disorders) | 55 | 6 | 33 | 9 | 2
PAIN (General disorders) | 16 | 5 | 5 | 3 | 2
PYREXIA (General disorders) | 77 | 7 | 56 | 21 | 4
CELLULITIS (Infections and infestations) | 13 | 3 | 7 | 0 | 0
LUNG INFECTION (Infections and infestations) | 1 | 0 | 3 | 3 | 0
NASOPHARYNGITIS (Infections and infestations) | 13 | 2 | 5 | 0 | 2
ORAL CANDIDIASIS (Infections and infestations) | 16 | 4 | 4 | 3 | 0
ORAL HERPES (Infections and infestations) | 15 | 2 | 8 | 6 | 0
PHARYNGITIS (Infections and infestations) | 9 | 1 | 5 | 1 | 2
PNEUMONIA (Infections and infestations) | 16 | 0 | 12 | 4 | 4
RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 2 | 4 | 0 | 0
SKIN INFECTION (Infections and infestations) | 5 | 0 | 0 | 1 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 | 1 | 5 | 1 | 1
URINARY TRACT INFECTION (Infections and infestations) | 16 | 3 | 14 | 0 | 2
CONTUSION (Injury, poisoning and procedural complications) | 16 | 3 | 7 | 2 | 2
FALL (Injury, poisoning and procedural complications) | 14 | 2 | 7 | 1 | 1
LACERATION (Injury, poisoning and procedural complications) | 3 | 0 | 2 | 0 | 2
WEIGHT DECREASED (Investigations) | 30 | 3 | 2 | 1 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 61 | 8 | 33 | 7 | 2
DEHYDRATION (Metabolism and nutrition disorders) | 11 | 2 | 4 | 1 | 0
FLUID OVERLOAD (Metabolism and nutrition disorders) | 8 | 2 | 0 | 3 | 0
FLUID RETENTION (Metabolism and nutrition disorders) | 5 | 0 | 0 | 3 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 11 | 1 | 11 | 7 | 1
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 16 | 0 | 6 | 3 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 54 | 6 | 45 | 16 | 3
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 21 | 2 | 9 | 6 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 9 | 0 | 12 | 3 | 1
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 19 | 2 | 8 | 6 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 33 | 2 | 11 | 3 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 36 | 5 | 22 | 2 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 12 | 2 | 4 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 21 | 2 | 3 | 1 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 26 | 2 | 11 | 2 | 2
ACUTE MYELOID LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 27 | 2 | 21 | 1 | 0
DIZZINESS (Nervous system disorders) | 42 | 3 | 15 | 4 | 1
HEADACHE (Nervous system disorders) | 31 | 1 | 19 | 6 | 3
SCIATICA (Nervous system disorders) | 4 | 2 | 2 | 0 | 0
AGITATION (Psychiatric disorders) | 6 | 3 | 3 | 0 | 1
ANXIETY (Psychiatric disorders) | 15 | 4 | 6 | 2 | 2
CONFUSIONAL STATE (Psychiatric disorders) | 14 | 3 | 8 | 3 | 1
INSOMNIA (Psychiatric disorders) | 36 | 2 | 11 | 4 | 1
HAEMATURIA (Renal and urinary disorders) | 5 | 3 | 8 | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 7 | 2 | 3 | 3 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 4 | 2 | 3 | 1 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 5 | 2 | 1 | 2 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 54 | 6 | 36 | 6 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 41 | 6 | 35 | 4 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 6 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 29 | 5 | 21 | 2 | 4
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 4 | 2 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 16 | 2 | 11 | 4 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 2 | 1 | 2
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 10 | 3 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 18 | 0 | 6 | 3 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 12 | 0 | 16 | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 25 | 1 | 10 | 6 | 0
RASH (Skin and subcutaneous tissue disorders) | 26 | 0 | 14 | 8 | 1
SKIN LESION (Skin and subcutaneous tissue disorders) | 4 | 2 | 5 | 0 | 1
SKIN ULCER (Skin and subcutaneous tissue disorders) | 7 | 2 | 2 | 1 | 0
HAEMATOMA (Vascular disorders) | 16 | 2 | 7 | 1 | 2
HYPERTENSION (Vascular disorders) | 16 | 1 | 13 | 4 | 2
HYPOTENSION (Vascular disorders) | 19 | 3 | 14 | 1 | 1
PHLEBITIS (Vascular disorders) | 7 | 2 | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator shall have the right to publish and/or present study data provided that the investigator shall (i) furnish the sponsor a copy of any proposed publication or presentation 60 days in advance of the submission and (ii) delete any confidential information of the sponsor and (iii) delay submission for up to 90 days to permit the preparation and filing of intellectual property applications or until sponsor gives its consent in a timely manner.